CLINICAL TRIAL: NCT06236399
Title: EEG Study of the Rhythmic Nature of Human Visual Perception and Attention
Brief Title: An EEG Study on the Rhythmic Nature of Perception and Attention
Status: Recruiting | Type: Observational
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Luca Ronconi, Professor, Università Vita-Salute San Raffaele
Other Study IDs: EEGVISION-01
Record Dates: First submitted 2024-01-08; First posted 2024-02-01 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Human Brain and Cognition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study involved healthy volunteers (n= 200), in a single center, low-risk intervention protocol of a non-profit nature. The objective of the study is to investigate the neural mechanisms of visual perception and attention, with particular reference to neural oscillations, in the general population through electroencephalogram (EEG) recording and the administration of simple visual tasks on a PC. The study presented is not associated with risks, as EEG is a non-invasive technique for which there are no known contraindications or adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 35 years
* able/willing to sign the informed consent
* normal or corrected-to-normal vision and hearing

Exclusion Criteria:

- history of severe/major neurological or psychiatric conditions

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy human volunteers
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-11-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Electroencephalographic (EEG) oscillatory amplitude | during the intervention
  Amplitude of EEG oscillations in theta, alpha and beta frequency bands
Electroencephalographic (EEG) oscillatory frequency | during the intervention
  Frequency of EEG oscillations in theta, alpha and beta frequency bands
Electroencephalographic (EEG) oscillatory phase coherence | during the intervention
  Phase coherence of EEG oscillations in theta, alpha and beta frequency bands
Autism Quotient (AQ) | during the intervention
  Personality questionnaire measuring subclinical autistic traits. Higher score mean worse outcome. Score range: min.= 0, max.= 50.
Schizotypal Personality Questionnaire (SPQ) | during the intervention
  Personality questionnaire measuring subclinical schizotypal traits. Higher score mean worse outcome. Score range: min.= 0, max.= 74.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy